CLINICAL TRIAL: NCT05973318
Title: An Open-label, Randomized, Controlled, Comparative Efficacy and Safety Study of Dorzotimol Eye Drops, 20 mg/mL + 5 mg/mL (JGL dd, Croatia), vs. Cosopt® Eye Drops, 20 mg/mL + 5 mg/mL (Merck Sharp & Dohme, France) in Patients With POAG
Brief Title: Comparative Study of Dorzotimol Eye Drops, 20 mg/mL + 5 mg/mL Versus Cosopt® Eye Drops, 20 mg/mL + 5 mg/mL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jadran Galenski laboratorij d.d. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DORZOTIMOL-10/2015
Record Dates: First submitted 2023-07-26; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Primary Open Angle Glaucoma of Both Eyes
Keywords: Glaucoma; Intraocular pressure; Treatment
MeSH Terms: conditions — Glaucoma | interventions — dorzolamide-timolol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with primary open-angle glaucoma receiving Dorzotimol eye drops, 20 mg/mL + 5 mg/mL (Experimental): Dosing schedule b.i.d., 12 weeks
  Interventions: Drug: Dorzotimol eye drops, 20 mg/mL + 5 mg/mL
- Patients with primary open-angle glaucoma receiving Cosopt eye drops, 20 mg/mL + 5 mg/mL (Active Comparator): Dosing schedule b.i.d., 12 weeks
  Interventions: Drug: Cosopt eye drops, 20 mg/mL + 5 mg/mL

INTERVENTIONS:
Drug: Dorzotimol eye drops, 20 mg/mL + 5 mg/mL — Dosing schedule b.i.d.
  Other Names: Dorzotimol
  Arms: Patients with primary open-angle glaucoma receiving Dorzotimol eye drops, 20 mg/mL + 5 mg/mL
Drug: Cosopt eye drops, 20 mg/mL + 5 mg/mL — Dosing schedule b.i.d.
  Other Names: Cosopt
  Arms: Patients with primary open-angle glaucoma receiving Cosopt eye drops, 20 mg/mL + 5 mg/mL

SUMMARY:
The goal of this study is to compare efficacy and safety of Dorzotimol eye drops, 20 mg/mL + 5 mg/mL manufactured by JADRAN-GALENSKI LABORATORIJ d.d. (Croatia) aimed at lowering elevated IOP in patients with ocular hypertension and primary open-angle glaucoma (POAG) versus Cosopt® eye drops, 20 mg/mL + 5 mg/mL manufactured by Laboratoires Merck Sharp & Dohme-Chibret, France. The main questions it aims to answer are:

* if the efficacy of the investigational drug and the reference drug in patients with ocular hypertension and primary open-angle glaucoma is equal;
* if the safety of the investigational drug and the reference drug in patients with ocular hypertension and primary open-angle glaucoma is equal.

A total of 110 participants were screened and randomized 1:1 to the investigational drug (Dorzotimol) group or the reference drug (Cosopt) group. 55 patients were recruited in each group.

Researchers compared the investigational drug (Dorzotimol) group with the reference drug (Cosopt) group to see if the efficacy and safety of the investigational drug and the reference drug in patients with ocular hypertension and primary open-angle glaucoma are equal.

DETAILED DESCRIPTION:
Study Title:

An open-label, randomized, controlled, comparative efficacy and safety study of Dorzotimol eye drops, 20 mg/mL + 5 mg/mL, manufacturer: JADRAN - GALENSKI LABORATORIJ d.d., Croatia, vs. Cosopt® eye drops, 20 mg/mL + 5 mg/mL, manufacturer: Laboratoires Merck Sharp & Dohme-Chibret, France, in patients with primary open-angle glaucoma.

Protocol No. DORZOTIMOL-10/2015, version No. 1.2 of 16.05.2017. RCT No. 632 of 09.09.2016.

Investigators:

1. Abdulaeva Elmira Abdulaevna (Test facility No.4)
2. Eryomina Alyona Victorovna (Test facility No.6)
3. Lisitsyn Alexey Borisovich (Test facility No.7)
4. Doga Alexander Victorovich (Test facility No.9)

Test facilities:

No.4. State autonomous healthcare institution 'Republican Clinical Ophthalmological Hospital of the Ministry of Health of the Republic of Tatarstan', 420012, Republic of Tatarstan, Kazan, Butlerova St., 14.

No.6. Federal state autonomous institution 'Acad. S.N. Fyodorov Eye Microsurgery Interbranch Science and Technology Complex', Ministry of Health of the Russian Federation, 127486, Moscow, Beskudnikovsky Blvd., 59A (branch: 630071, Novosibirsk, Kolkhidskaya St., 10).

No.7. State healthcare institution of Yaroslavl region 'Clinical Hospital No. 8', 150030, Yaroslavl, Suzdalskoe Highway, 39.

No.9. Federal state autonomous institution 'Acad. S.N. Fyodorov Eye Microsurgery Interbranch Science and Technology Complex', Ministry of Health of the Russian Federation, 127486, Moscow, Beskudnikovsky Blvd., 59A

Study period:

First patient enrollment date: 10 April 2017 Study completion date: 17 September 2018

Phase:

III (a safety and efficacy study)

Study objective:

The study objective was to evaluate the efficacy and safety of Dorzotimol eye drops, 20 mg/mL + 5 mg/mL, manufacturer: JADRAN - GALENSKI LABORATORIJ d.d., Croatia, designed to reduce elevated intraocular pressure in patients with primary open-angle glaucoma (POAG), vs. Cosopt® eye drops, 20 mg/mL + 5 mg/mL, manufacturer: Laboratoires Merck Sharp & Dohme-Chibret, France.

Study tasks:

* Demonstrate sufficient similarity of the efficacy profiles of the test and reference product in patients with primary open-angle glaucoma.
* Demonstrate sufficient similarity of the safety profiles of the test and reference product in patients with primary open-angle glaucoma.

Study design:

A multicenter, prospective, open-label, randomized, comparative, controlled, parallel-arm study evaluating the efficacy and safety in patients with a specific disease.

Study subjects: 110 patients (55 patients in each group) with elevated intraocular pressure induced by primary open-angle glaucoma (POAG), males and females in the age bracket of 18 to 75 years conforming to the inclusion/exclusion criteria.

Patients randomized: 110 Dropouts: 0 Per protocol population: 110 Safety population: 110 Drug therapy type

Test product:

Trade name: Dorzotimol INN or generic name: dorzolamide+timolol Pharmaceutical form: eye drops

Composition per 1 mL:

Active ingredients: dorzolamide hydrochloride 22.25 mg (equivalent to dorzolamide 20 mg), timolol maleate 6.83 mg (equivalent to timolol 5 mg).

Excipients: benzalkonium chloride (as 50% solution), mannitol, sodium citrate, sodium hydroxide, hydroxyethyl cellulose, purified water.

Manufacturer: JADRAN - GALENSKI LABORATORIJ d.d., Croatia Posology and method of administration: Instillation into the conjunctival sac of 1 drop twice daily for 12 weeks.

Reference product description and labeling:

Trade name: Cosopt® INN or generic name: dorzolamide+timolol Pharmaceutical form: eye drops

Composition:

Active ingredients: dorzolamide 20 mg (dorzolamide hydrochloride 22.26 mg) and timolol 5 mg (timolol maleate 6.83 mg).

Excipients: benzalkonium chloride (as 50% benzalkonium chloride solution) 0.075 mg (0.15 mg), sodium citrate 2.94 mg, mannitol 16.00 mg, hyetellose (hydroxyethyl cellulose) 4.75 mg, 1M sodium hydroxide solution q.s. to рН 5.6, water for injection q.s. to 1 mL.

Manufacturer: Laboratoires Merck Sharp & Dohme-Chibret, France Study duration: Screening: 7 days. Washout period: 7 days. The comparison product treatment lasted for 12 weeks (84±2 days), which was consistent with the reference product PIL. Follow-up period for safety evaluation: 7 days. The overall study duration per patient did not exceed 100 days.

The efficacy was established based on analysis of the parameters as follows:

Primary endpoint

* Mean IOP change from baseline. Secondary endpoints
* IOP reduction rate to the target level of ≤ 18 mm Hg.
* IOP reduction rate greater than 20%.
* IOP reduction rate greater than 30%. Safety evaluation
* Incidence of other adverse events to a greater or lesser extent linked to the test or reference product, including those evaluated from laboratory test findings.
* Treatment safety will be assessed from recording adverse events via analysis of complaints and symptoms, evaluation, and interpretation of the findings of instrumental monitoring (biomicroscopy, ophthalmoscopy, IOP measures, perimetry) and laboratory tests.
* Given that the test product may cause miosis resulting in transient visual acuity reduced, the contribution of the visual acuity parameter 'Vis' is not taken into account when assessing the treatment success.

Statistical analysis Statistical analysis was performed using Statsoft Statistica Professional 13 and Microsoft Excel 2016 software.

The Shapiro-Wilk test was used to evaluate the normality of distribution of quantitative attributes. Parametric tests were used for testing statistical hypotheses for parameters with the normal distribution, whereas nonparametric tests were used for parameters with the variance of the distribution. Student's t-test and Mann-Whitney U test were used for comparing the study groups in terms of quantitative attributes. The comparison of intragroup parameters before and after treatment was performed using the dependent samples t-test or the Wilcoxon test. The intragroup comparisons were also performed using nonparametric repeated measures ANOVA (the Friedman test). Qualitative attributes were analyzed using Pearson's χ2 test or Fisher's exact test (if the attribute incidence rate in at least one subgroup was ≤ 5).

Statistically significant are differences with p-values < 0.05. Efficacy analysis of the comparison products provides for a conclusion on

• Noninferiority of the test product Dorzotimol, eye drops (JADRAN - GALENSKI LABORATORIJ d.d., Croatia) vs. reference product Cosopt®, eye drops (Laboratoires Merck Sharp & Dohme-Chibret, France) by the primary endpoint:

* No statistically significant intergroup differences have been observed regarding a mean intraocular pressure change from baseline either in the treatment or control group (p = 0.0939; Mann-Whitney U test).
* The efficacy differences between the test and reference product by the primary criterion do not exceed the noninferiority margin of 1.5 mm Hg.

Intergroup efficacy comparisons of the comparison products by the secondary endpoints have also been performed, with statistical significance of intergroup differences evaluated:

* No statistically significant intergroup differences have been observed regarding the IOP reduction rate to the target level of ≤ 18 mm Hg either in the treatment or control group (p = 0.3061; Pearson's χ2 test), which is indicative of Dorzotimol noninferiority by this parameter vs. reference product.
* No statistically significant intergroup differences have been observed regarding the IOP reduction rate greater than 20% at visit 6 from baseline either in the treatment or control group (p = 0.6336; Pearson's χ2 test), which is indicative of Dorzotimol noninferiority by this parameter vs. reference product.
* No statistically significant intergroup differences have been observed regarding the IOP reduction rate greater than 30% at visit 6 from baseline either in the treatment or control group (p = 0.4492, Pearson's χ2 test), which is indicative of Dorzotimol noninferiority by this parameter vs. reference product.

The product safety was assessed from the vital parameters evaluation results, laboratory test and instrumental monitoring data as well as the adverse event occurrence and severity.

The safety evaluation provided for the conclusions as follows:

* Analysis of these AEs is indicative of comparable safety of the test product:

  * AE occurrence in the treatment group does not differ reliably from AE occurrence in the control group (p = 0.3242; Pearson's χ2 test).
  * AE link to the test product was most characterized as 'probable'; there were no statistically significant intergroup differences by this parameter either (p = 0.2774).
  * AE severity was most characterized as mild; there were no statistically significant intergroup differences by this parameter either (p = 0.4309).
* There were no statistically significant intergroup differences either when assessing physical examination parameters or in terms of individual dynamics level.
* Analysis of the patients' laboratory test findings has identified statistically reliable differences by certain parameters (hemoglobin, glucose levels); however, these differences are also linked to patients' personality traits.

Thus, based on all criteria specified in the Clinical Trial Protocol, the test product Dorzotimol and reference product Cosopt® demonstrate close efficacy and safety parameters. There are no statistically significant intergroup differences by any efficacy criteria tested. The efficacy differences between the test and reference product by the primary criterion do not exceed the noninferiority margin of 1.5 mm Hg. The above-stated provides for a conclusion on the test product Dorzotimol noninferiority vs. reference product Cosopt®.

ELIGIBILITY:
Inclusion Criteria:

* Females or males in the age bracket of 18 to 75 years.
* Established stage I and II primary open-angle glaucoma in one or both eyes.
* Intraocular pressure (IOP) level: 22-36 mm Hg (by Goldmann applanation tonometry).
* Visual acuity 0.3 or better on the tested eye.
* Taking topical prostaglandin analogs as monotherapy at least 3 months prior to the enrollment into the study and poor IOP control (> 21 mm Hg) or failure to achieve the target IOP, as estimated by the physician.
* Patients who have signed an informed consent to participate in the study.
* For females of child-bearing potential - a negative pregnancy test and consent to use reliable contraception methods throughout the study

Exclusion Criteria:• Contraindications or hypersensitivity to the active ingredients (dorzolamide and/or timolol) or excipients.

* The only eye.
* Visual acuity ˂ 0.3 after correction.
* An active infectious inflammatory process on the tested eye within 3 months prior to pre-study medical examination.
* Pronounced visual field defects (III and IV stage open-angle glaucoma).
* IOP > 36 mm Hg or < 22 mm Hg as at the IOP measuring at 11:00 a.m. (±1 h) in any of the eyes on the screening visit day.
* Closed or nearly closed anterior chamber angle (ACA) or history of acute angle close.
* Surgical and laser eye interventions over the last 3 months.
* Manifest ocular media opacification hindering the treatment efficacy evaluation.
* Other eye diseases that may affect dynamics of the parameters used for the treatment efficacy evaluation.
* Inflammatory conditions of the eye and appendages (blepharitis, conjunctivitis).
* Corneal dystrophies.
* The patient's participation in another clinical trial for the last 3 months.
* Sinus bradycardia.
* Second-degree and third-degree AV block.
* Cardiogenic shock.
* Decompensated cardiovascular diseases (angina pectoris > functional class II, arterial hypertension [systolic pressure > 140 mm Hg, diastolic pressure > 90 mm Hg]), apparent heart failure.
* Severe renal failure (CC < 30 mL/min).
* Airway hyperresponsiveness, bronchial asthma, history of bronchial asthma, severe chronic obstructive pulmonary disease.
* Any other systemic or mental disorder/condition (unmanageable arterial hypertension, decompensated diabetes mellitus, severe renal impairment, hyperchloremic acidosis) or clinically relevant abnormal laboratory tests at screening that, in the Investigator's opinion, may put a patient to a significant risk, or compromise the study results, or appreciably affect the possibility for the patient to participate in the study.
* A patient who is unlikely to comply with the protocol requirements, e.g., is undisposed to cooperation, and is unlikely to complete the study.
* Females and males of reproductive age refusing to use efficacious contraception methods.
* Females during pregnancy and breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-09-17 (Actual)

PRIMARY OUTCOMES:
Mean IOP change from baseline | 12 weeks
  Mean IOP change from baseline on visit 5 comparing with visit 0

SECONDARY OUTCOMES:
IOP reduction rate to the target level of ≤ 18 mm Hg | 12 weeks
  IOP reduction rate to the target level of ≤ 18 mm Hg on visit 5 comparing with visit 0
IOP reduction rate greater than 20% | 12 weeks
  IOP reduction rate greater than 20% on visit 5 comparing with visit 0
IOP reduction rate greater than 30% | 12 weeks
  IOP reduction rate greater than 30% on visit 5 comparing with visit 0

CONTACTS AND LOCATIONS:
Overall Officials: Elmira Abdulaeva, Principal Investigator — Republican Clinical Ophthalmological Hospital of the Ministry of Health of the Republic of Tatarstan
Locations (1):
- Republican Clinical Ophthalmological Hospital of the Ministry of Health of the Republic of Tatarstan, Kazan', Russia

IPD SHARING:
Plan to Share IPD: No